CLINICAL TRIAL: NCT01802762
Title: A New Multi-parameter Neuromonitoring System to Save Patients' Lives in Stroke and Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeMoDevices AG (Industry)
Collaborators: Medical University of Graz (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-1.000_NeMo_C001 / MUG; E!6526_OPTO-BRAIN (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2013-02-24; First posted 2013-03-01 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Subarachnoid Hemorrhage; Optical Imaging
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeMo Patch and NeMo Probe (Other): TBI and SAH patients, one arm
  Interventions: Device: NeMo Patch and NeMo Probe

INTERVENTIONS:
Device: NeMo Patch and NeMo Probe — A plaster based patch (NeMo Patch) and a combined probe for ICP monitoring and near infrared spectroscopy (NIRS) are applied as sensors. Data are collected by a NIRS instrument (NeMo Control Unit)

SUMMARY:
To assess the feasibility of a new neuromonitoring system (NeMoSystem including NeMo Probe and NeMo Patch) and the accuracy of the measurement values (cerebral blood flow (CBF); cerebral blood volume (CBV)) obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patient, ≥ 18 and ≤ 75 years
2. Patient with severe SAH (GCS ≤ 12) or severe TBI (GCS ≤ 8)
3. Decreased level of consciousness with the need for ICP monitoring for an estimated duration of more than 3 days
4. Negative pre-treatment serum pregnancy test for female patients with childbearing potential
5. In patients with severe SAH or severe TBI with need for ICP monitoring an acute emergency situation exists. The inclusion follows

Exclusion Criteria:

1. Known kidney disease, defined as plasma creatinine > 120 µmol/l
2. Known liver disease, defined as GOT > 200U/l
3. History of allergic disorders, including allergic reactions against contrast agents containing iodine, against ICG and against plasters, as well as patients with thyroid disease causing hyperthyroidism
4. Pre-existing disability and/or legal representative
5. Participation in another interventional clinical trial within the last 30 days before start of treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of the neuromonitoring system and the accuracy of the measurement values. | Day 28 after removal of medical device
  Feasibility:
  User acceptance: For NeMo Probes in comparison to conventional probes for intracranial pressure (ICP-) monitoring; for NeMo Patch in comparison to patches for electroencephalography (EEG) monitoring.
  Detailled evaluation of user acceptance:
  * Incidence of concerns of users in relation to the installation, function and removal of the NeMo System (= NeMo Probe, NeMo Patch, NeMo Control Unit and NeMo Software pre-installed on a Medical PC)
  * User-friendliness with a 3-graded scale (equal, better, worse) compared to conventional devices
  Accuracy of measurements:
  -Patients: Results from repeated measurements of mean transit time of ICG (mttICG), cerebral blood flow (CBF) and cerebral blood volume (CBV)
  Safety parameters:
  Incidence of complications (infections, brain tissue damage, haemorrhage) compared to historical series (patches for EEG and for BIS measurements; conventional probes for ICP monitoring)

SECONDARY OUTCOMES:
To demonstrate the ability of the neuromonitoring system to detect secondary ischemic events in patients with severe subarachnoid haemorrhage (SAH) or severe traumatic brain injury (TBI). | Day 28 after removal of medical device
  Results concerning sensitivity and specificity to detect symptomatic vasospasm in patients with subarachnoid hemorrhage (SAH) (correlation of events with CBF values < 15 ml/100g/min with defined criteria for vasospasm) Results concerning sensitivity and specificity to detect secondary infarctions and critical ICP values in TBI patients (correlation of events with CBF values < 15 ml/100g/min with defined criteria for secondary infarction) Results from repeated measurements for the difference between measurement values obtained with the NeMo Patch and the NeMo Probe, quantified with mathematical models

CONTACTS AND LOCATIONS:
Locations (2):
- Dept. of Neurosurgery, Medical University of Graz, Graz, Austria
- Neurointensive Care Unit, University Hospital Zurich, Zurich, Switzerland